CLINICAL TRIAL: NCT06032949
Title: Vialize Use for the Reduction of Vascular Groin Incisional Dehiscence and Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202301216
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Vascular Diseases
Keywords: groin infections; quality of life; readmission; groin incisions
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients from 2 populations will be included: high-risk patients (any of the following: redo groin incision, active smoker, A1c >/= 9.0, BMI >/= 30) and non-high-risk patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vialize (Other): Vialize is a lyophilized dehydrated complete human placental membrane allograft.
  Interventions: Other: Vialize

INTERVENTIONS:
Other: Vialize — Any patients undergoing surgeries involving a groin incision (e.g., femoropopliteal bypass, aortofemoral bypass, loop thigh graft, femoral exposure for delivery of device) will receive Vialize subcutaneously.

SUMMARY:
Groin incisions in vascular surgery have complications in up to 30% of cases at 30 days, resulting in reductions in patient quality of life and increased costs. Prior attempts at reducing this complication rate have been largely unsuccessful. The purpose of this study is to determine the feasibility of routine Vialize use for vascular surgeries involving a groin incision and to determine the rates of surgical site infection/dehiscence in such patients receiving subcutaneous Vialize.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of patients undergoing vascular procedures with groin incisions. Patients must be at least 18- years-old and able to complete baseline measurements. All subjects will be compensated. Patients undergoing treatment for peripheral arterial disease (e.g., femoropopliteal bypass), aneurysm disease (e.g., aortofemoral bypass), end-stage kidney disease (e.g., loop thigh graft), and miscellaneous procedures (e.g., femoral exposure for delivery of device) will be eligible.

Exclusion Criteria:

* Patients undergoing use of negative pressure wound therapy (e.g., Prevena) and local antibiotic placement (e.g., vancomycin powder) will be excluded. Additionally, organ-transplant recipients will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
The rate of infection at 90-day post-op follow-up in patients receiving Vialize during vascular surgeries involving a groin incision. | 90-day post-op follow-up
  Aim 1

SECONDARY OUTCOMES:
The patient quality of life (EQ-5D) | 90-day post-op follow-up
return to OR for groin infection | 90-day post-op follow-up
Readmission or prolongation of the index admission for groin infection | 90-day post-op follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Samir Shah, MD, MPH, Principal Investigator — COLLEGE-MEDICINE MD-SURGERY MD-SURGERY-VASCULAR
Locations (1):
- UF Health Heart & Vascular Hospital, Gainesville, Florida, United States